CLINICAL TRIAL: NCT01320462
Title: Smoking Cessation Program in the Preadmission Clinic:The Combination of Counseling, Pharmacotherapy and Quit Line
Brief Title: Smoking Cessation Program in the Preadmission Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Frances Chung, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WS836526
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2016-06

CONDITIONS: Smoking
Keywords: Smoking; quit; surgery; anesthesia; champix
MeSH Terms: conditions — Smoking | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking cessation group (Experimental): Counselling, Pharmacotherapy and Smokers Help Line
  Interventions: Drug: Smoking cessation counselling group
- Control group (Other): Brief informatin about quitting and smokers help line
  Interventions: Other: Control group:

INTERVENTIONS:
Drug: Smoking cessation counselling group — The smoking-cessation program has three components; structured preoperative counseling, pharmacotherapy with varenicline for three months, and referral to the quit line (Smokers' Helpline) for proactive telephone counseling and follow up
  Arms: Smoking cessation group
Other: Control group: — Interventions in the control group will be a brief advice regarding smoking cessation and provision of the quit line's information.
  Arms: Control group

SUMMARY:
Main Hypothesis: The multifaceted intervention (preoperative counseling, pharmacotherapy by varenicline and follow up by quit line) in the preoperative clinic is more effective than the simple preoperative smoking intervention (brief advice and provision of information about the quit lines ) in terms of short-term and long-term quit rates

Objectives: To evaluate the effectiveness and feasibility of a multifaceted intervention (preoperative counseling, pharmacotherapy by varenicline and follow up by the quit line) in the preoperative clinic to help surgical patients quit smoking perioperatively and for the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Patients who smoke more than 10 cigarettes per day for more than 1 year
* And had no period of smoking abstinence longer than 3 months in the past year.
* Patients who are scheduled to have any elective surgery next 7 to 60 days. Patients > 18 years of age

Exclusion Criteria:

* Patients unwilling or unable to give informed consent
* Patients who are pregnant and breast feeding
* Patients with any psychiatric disorder
* Patients who used nicotine replacement / bupropion within previous 3 months
* Cardiovascular disease within the past 6 months
* Any serious or unstable disease within the past 6 months
* Drug or alcohol abuse within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2010-12; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
pre-surgery counseling for quit smoking | 1 year after surgery
  In order to determine the prevalence of abstinence in long-term follow up (4, 12, 24 and 52 weeks), patients will be asked the following questions:
  * Have you been abstinent from smoking for the past four weeks? (4-week abstinence)
  * Do you currently smoke cigarettes everyday? (point prevalence)
  * Have you been abstinent from smoking since the last time you quit smoking? (continuous abstinence)

SECONDARY OUTCOMES:
perioperative complications | 3 months after surgery
  Secondary outcome measures that will be studied are as follows: The changes in the number of cigarettes consumed per day or 'stage of change' at 4, 12, 24 and 52 weeks after the initial assigned target quit date. The incidence of perioperative complications (until 30 days after surgery) as well as medication-related adverse events (and serious adverse events) will also be recorded (only those who in the smoking-cessation program).

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto Western Hospital, Department of Aneshtesia, Toronto, Ontario
  - Mount Sinai Hospital, Department of Anesthesia, Toronto, Ontario